## Response to inflammatory challenge in major depressive disorder

Protocol #2016-002-03

NCT03142919

10/12/2017

Data will be analyzed using linear mixed models with group (high versus low-CRP) and drug (LPS versus saline) as between subject factors, and time as the within-subject factor; the fixed-effects also include their 2-and 3-way interactions. Within-subject dependency will be captured by random subject intercepts and/or random time slopes. The need for random slopes and the addition of age, self-reported sex, BMI, and medication status (unmedicated versus medicated) as covariates will be evaluated by Bayesian Information Content. Where appropriate, data will be normalized to z-scores using the ordered quantile method and effect sizes will be calculated by converting the F- and t-statistics into (partial)  $\eta$ ! and Cohen's d. F- and t-tests are one- and two-tailed, respectively. The analyses will be conducted with R programming language (version 4.3.1) using bestNormalize (version 1.9.1), ImerTest (version 3.1.3), and emmeans (version 1.8.8) packages for data normalization, linear mixed-effects models, and post hoc comparisons.